CLINICAL TRIAL: NCT05863689
Title: Microvascular Ocular Changes of Systemic Lupus Erythematous
Acronym: VascLup
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar Universitário de Santo António (Other)
Responsible Party: Sponsor
Other Study IDs: VascLup
Record Dates: First submitted 2023-04-28; First posted 2023-05-18 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-04

CONDITIONS: Eye Manifestations; Lupus Erythematosus, Systemic
MeSH Terms: conditions — Eye Manifestations; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SLE Patients: Patients fulfilling the 1997 revised American College of Rheumatology (ACR) criteria for the diagnosis of SLE (21) and aged between 18 and 80 years old.
  Ophthalmological inclusion criteria: (1) best-corrected visual acuity ≤ 0.3 LogMAR, (2) intra-ocular pressure <21 mm Hg on diurnal testing with measurements using Goldmann applanation tonometry, (3) spherical equivalent refractive error between -6.0 and +4.0 diopters, and (4) open anterior chamber angle on slit lamp examination.
  Interventions: Diagnostic Test: Spectralis SD-OCT
- Healthy Controls: Healthy controls matched for sex and age with SLE Patients. Ophthalmological inclusion criteria: (1) best-corrected visual acuity ≤ 0.3 LogMAR, (2) intra-ocular pressure <21 mm Hg on diurnal testing with measurements using Goldmann applanation tonometry, (3) spherical equivalent refractive error between -6.0 and +4.0 diopters, and (4) open anterior chamber angle on slit lamp examination.
  Interventions: Diagnostic Test: Spectralis SD-OCT

INTERVENTIONS:
Diagnostic Test: Spectralis SD-OCT — Optical Coherence Tomography

SUMMARY:
The goal of this observational study is to to assess the ocular microvascular status of SLE patients with inactive disease and without ocular involvement. The main questions it aims to answer are:

* the choroidal vascular status and thickness in SLE
* the retinal macular microvascular status and structure in SLE

Participants will be assessed with Spectral Domain Optical Coherence Tomography (SD-OCT). Researchers will compare SLE patients with healthy controls matched for age and sex.

DETAILED DESCRIPTION:
The investigators will perform a cross-sectional evaluation of 25 SLE patients and 25 healthy controls matched for sex and age, using a Spectral Domain Optical Coherence Tomography (SD-OCT) with Enhanced Depth Imaging for choroidal assessment and with Angiography module to assess the retinal and choriocapillaris vasculature. Processing of image with external software will be performed to calculate the main outcomes: retinal vessel density, foveal avascular zone parameters and the choroidal vascular index.

ELIGIBILITY:
Systemic inclusion criteria for SLE patients:

* fulfill the 2019 European League Against Rheumatism (EULAR) / American College of Rheumatology (ACR) classification criteria for the diagnosis of SLE
* age between 18 and 80 years
* no disease activity (SLEDAI <3)
* no risk factors for drug toxicity

Systemic inclusion criteria for control group:

* no systemic diseases
* age between 18 and 80 years

Systemic exclusion criteria:

* arterial hypertension (defined as systolic blood pressure higher than 140 mm Hg or diastolic blood pressure higher than 90 mm Hg) or medically treatment for hypertension
* diabetes mellitus
* nephropathy or other documented microvascular complications
* secondary Sjögren syndrome
* local or systemic inflammatory diseases (other than SLE)
* smokers of more than 20 cigarettes a day
* pregnancy.

Ophthalmological inclusion criteria:

* best-corrected visual acuity ≤ 0.3 LogMAR
* intra-ocular pressure <21 mm Hg on diurnal testing with measurements using Goldmann applanation tonometry
* spherical equivalent refractive error between -6.0 and +4.0 diopters
* open anterior chamber angle on slit lamp examination.

Ophthalmic exclusion criteria:

* established primary ocular diseases including a history of any retinal or optic nerve disease
* presence of significant lens opacities (Lens Opacities Classification System III equal to or more stage 2)
* retinopathy
* high refractive error
* ocular hypertension
* previous intraocular surgery or trauma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients fulfilling the 2019 European League Against Rheumatism (EULAR) / American College of Rheumatology (ACR) classification criteria for the diagnosis of SLE and aged between 18 and 80 years old and an age and sex-matched group of healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of retinal vessel density | 6 months
  Comparison of retinal vessel density of superficial and deep plexuses between SLE patients and healthy controls using OCT Angiography.
Measurement of choroidal vascular index | 6 months
  Comparison of choroidal vascular index between SLE patients and healthy controls using OCT with Enhance Depth Imaging

CONTACTS AND LOCATIONS:
Overall Officials: André Ferreira, MD PhDc, Principal Investigator — Centro Hospitalar Universitário de Santo António
Locations (1):
- Centro Hospitalar Universitário de Santo António, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferreira A, Viveiros L, Faria R, Braganca F, Abreu AC, Santos D, Furtado MJ, Lume M, Meneres P, Andrade JP. Retinal microvascular changes in systemic lupus erythematosus assessed by optical coherence tomography angiography. Int J Retina Vitreous. 2024 Dec 18;10(1):94. doi: 10.1186/s40942-024-00617-6. PMID 39696716